CLINICAL TRIAL: NCT00542113
Title: Diabetes Virtual Trek Prevention: Obesity and Diabetes Prevention Through Science Enrichment
Brief Title: Diabetes Virtual Trek: Obesity and Diabetes Prevention Through Science Enrichment
Acronym: DvtENERGY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: Poudre School District, Fort Collins, CO (Unknown); Montezuma-Cortez School District, Cortez, CO (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H 00-301H R25 015646; R25RR015646 (NIH); R25RR020469 (NIH)
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: Parental; Parents; Prevention; Energy balance; Glucose regulation; Healthy lifestyles; Healthy families; Active living
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Parents of elementary school children in grades 2-6 participating in Program ENERGY -Intervention 1
  Interventions: Behavioral: DvtProgram ENERGY
- 2 (Experimental): Parents of elementary school children in grades 2-6 participating in Program ENERGY -Intervention 2
  Interventions: Behavioral: DvtProgram ENERGY
- 3 (Sham Comparator): Parents of elementary school children in grades 2-6 participating in Program ENERGY matched to the intervention groups
  Interventions: Behavioral: DvtProgramENERGY

INTERVENTIONS:
Behavioral: DvtProgram ENERGY — 11 - weekly or biweekly newsletters about diabetes and its prevention and family challenges sent home with children
  Arms: 2
Behavioral: DvtProgram ENERGY — 6 - weekly or biweekly newsletters about diabetes and its prevention and family challenges sent home with children
  Arms: 1
Behavioral: DvtProgramENERGY — Children participating in Program ENERGY but no newsletters or family challenges sent home to parents
  Arms: 3

SUMMARY:
The purpose of this study was to evaluate the effectiveness of a school-to-home education program for it's ability to increase knowledge about, and ability to prevent type two diabetes in children and parents.

DETAILED DESCRIPTION:
The study involved pre and post testing of parent's knowledge and behaviors relating to the prevention of type two diabetes, before and after a school based intervention designed to encourage school to home communication. Parents/Guardians and children, grades 2-6, from schools with high Hispanic enrollment during the 2001-2005 school year were used for both comparison and intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* Elementary school children in grade 2-6 in intervention or comparison classes/schools

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1703 (Actual)
Dates: Start 2001-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Diabetes knowledge and prevention of parents of elementary school children | one-three school year(s)

SECONDARY OUTCOMES:
Self-reported parental physical activity | one -three school year(s)

CONTACTS AND LOCATIONS:
Overall Officials: L. Arthur Campfield, PhD, Principal Investigator — Colorado State University
Locations (2):
- United States (2):
  - Montezuma-Cortez School District, Cortez, Colorado
  - Putnam, Tavelli, Bennett and Dunn Elementary Schools, Fort Collins, Colorado

REFERENCES:
- See also: Program ENERGY website — http://ProgramENERGY.org